CLINICAL TRIAL: NCT04318171
Title: The Evaluation of Tomographic 3D Ultrasound for the Assessment of Vascular Pathology
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20HH5799
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Carotid Artery Plaque
MeSH Terms: conditions — Carotid Stenosis | interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Carotid arteries.: No intervention is required. Routine Doppler assessment + 3D scan immediately afterwards.
  Interventions: Device: 3D Imaging.
- Peripheral arteries.: No intervention is required. Routine Doppler assessment + 3D scan immediately afterwards.
  Interventions: Device: 3D Imaging.
- AVF.: No intervention is required. Routine Doppler assessment + 3D scan immediately afterwards.
  Interventions: Device: 3D Imaging.
- Vein mapping: No intervention is required. Routine Doppler assessment + 3D scan immediately afterwards.
  Interventions: Device: 3D Imaging.

INTERVENTIONS:
Device: 3D Imaging. — When the normal Doppler assessment is done following nationally approved protocol for scanning Carotid arteries, lower and upper limb arteries, AVF and Vein mapping. PIUR tUS infinity system 3D Bluetooth motion sensor which is linked to video transmission box will be used to scan the patient's common carotid artery (CCA), internal carotid artery (ICA) and external carotid artery (ECA) in transverse view to obtain the following measurements:
  * Plaque volume where detectable.
  * Max area stenosis.
  * Volumetric stenosis.
  * Measured length.
  * 3D GSM. The entire assessment should not take more than 45 minutes.

SUMMARY:
This study concentrates on providing more ultrasound image details when scanning vascular system including arterial and venous systems.

A new sensor which provides 3D images is newly designed. It will be used in this study to find out whether it can change the future of vascular imaging or not.

DETAILED DESCRIPTION:
Ultrasound is ideal for diagnosing vascular pathology due to its advantage of using different elements within its transducers, such as beam steering, focusing and high frame rate. It is also available and low costs when compared to other diagnostic modalities such as Computed Tomography (CT scan) and Magnetic Resonance Imaging (MRI). In addition to that, Duplex ultrasound (DUS) uses high sound waves with no ionising radiation. Therefore, it's fairly safe to the patient with long term surveillance.

DUS provides valuable information in diagnosing vascular disease due to its ability to detect flow motion within a vessel. It is, therefore, able to define whether the vessel being scanned is narrowed, diseased or blocked.

3D Ultrasound: 3D ultrasound provides images from different angles for better detection of structures being assessed. Therefore, the accuracy of the vessels and anatomical structures around is high. 3D Volume now becomes available and can be calculated and potentially benefits patients by detecting and defining those who are at risk of vascular disease.

There are three types of 3D ultrasound which are:

* Mechanical 3D
* 3D and 4D matrix scanning.
* Freehand 3D sensor. (Will be used in this project).

The targeted structures are:

Carotid arteries. Peripheral arteries including upper and lower limbs. Arteriovenous Fistula. Vein mapping pre coronary artery bypass graft (CABG).

Carotid Plaque Volume:

In 2009, a joint working coordinated efforts between the United Kingdom (UK) Vascular Societies concurred that the North American Symptomatic Carotid Endarterectomy Trial (NASCET) method for evaluating and grading carotid artery disease should be utilised in the UK.

In addition to current criteria used for grading carotid stenosis, Carotid plaque volume (CPV) is a measurement that may be a better predictive of embolic risk and stroke. CPV may be used to determine whether the patients with <70% stenosis and large plaque volume are at risk as other patients who present with >70% focal and short stenosis. A significant benefit of measuring Carotid plaque volume is observing the progression or regression of the area affected. This can be done clinically and in a quite relevant time frame.

Peripheral arterial disease (PAD):

20% of patients aged < 60 are likely to suffer from PAD including those present with intermittent claudication and also patients with critical limb ischemia (5-10%) of cases).

Uncontrolled diabetes mellitus can lead to the diabetic foot which can cause further complications such as infection, ulcer and neuropathy. DUS plays a vital role in diagnosing PAD particularly for those who are unable to be investigated by other modalities. Until now, there has been no work or research done on assessing PAD plaque volume. Investigating PAD using 3D may give an accurate diagnosis and provide more image details which can lead to a better treatment plan either by using endovascular or surgical procedures.

Arteriovenous Fistula AVF:

DUS pre and post AVF is considered the golden method of mapping and routinely assessing AVF. Renal association guidelines has stated that patients should undergo DUS for mapping in particular for those who have had previous central vein catheterisation procedures.

DUS mapping has been proven that it can positively reduce surgical complications including immediate failure. DUS also provides valuable details on AVF function and complications post creation based on current criteria including inflow and outflow volume rate. In this research, 3D US will be used to determine whether it can provide better result in compare to DUS which is currently the most widely used imaging modality.

Vein mapping:

DUS is currently used as a gold standard for vein mapping prior CABG and provides sufficient details about saphenous veins patency and suitability for using them as autogenous graft 195. 3D US may provide better image quality in demonstrating small vein branches and may improve surgical outcomes by providing more details prior to harvesting. It may also provide better details for surgeons on where to make an incision and defining the best segment of the vain is much appropriate.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years age with vascular disease.
* Male / Female.

Exclusion Criteria:

* <18 years age.
* Patient with congenital vascular abnormalities/syndromes.
* Pregnant patients will not be recruited in this study. Patient's pregnancy status will be assessed on initial enrollment to exclude them from the study.
* Those unable to provide consent.
* Anyone who is taking part in any other research.
* Potential participants who might not adequately understand verbal explanations or written information given in English, or who have special communication needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients selected for this study must have arterial stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Peck systolic velocity | 12 weeks
  Normal peck systolic velocity (PSV) is 125cm/s. More than 250 cm/s considered 50% stenosis .
Peck systolic ration | 12 weeks
  Normal peak systolic velocity rations less than 1.5 and more than 2 is considered 50% stenosis. This can be calculated by measuring the peak systolic velocity within the stenotic area divided by either pre or post stenotic area.
Diameter reduction measurement | 12 weeks
  The ultrasound medicine does calculate the diameter reduction automatically when the operator places the calliper at the vessels wall.

SECONDARY OUTCOMES:
Plaque volume | 12 weeks
  3D laptop calculates the plaque volume automatically.
Max area stenosis. | 12 weeks
  3D laptop calculates the plaque volume automatically.
Volumetric stenosis. | 12 weeks
  3D laptop calculates the plaque volume automatically.
Measured length. | 12 weeks
  3D laptop calculates the plaque volume automatically.
3D GSM. | 12 weeks
  3D laptop calculates the plaque volume automatically.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No